CLINICAL TRIAL: NCT01019265
Title: A Randomised Open Label Parallel Group Study Comparing Norspan Patch and Oral Tramadol
Brief Title: A Study Comparing Norspan Patch and Oral Tramadol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mundipharma Korea Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BUP07-KR-001
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Osteoarthritis
Keywords: Norspan patch; Buprenorphine transdermal patch (BTDS); efficacy; buprenorphine
MeSH Terms: conditions — Osteoarthritis | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Norspan patch (Buprenorphine TDS) (Experimental)
  Interventions: Drug: Buprenorphine 5mg, 10mg, 20mg vs Tramadol 100mg
- TramadolSR tab (Tridol SR tab) (Active Comparator)
  Interventions: Drug: Buprenorphine 5mg, 10mg, 20mg vs Tramadol 100mg

INTERVENTIONS:
Drug: Buprenorphine 5mg, 10mg, 20mg vs Tramadol 100mg — Comparing pain intensity between intervention drugs (Norspan® and Tridol®)
  Other Names: Norspan patch; Buprenorphine transdermal system (BTDS)

SUMMARY:
This trial was designed for comparison and evaluation of the efficacy and safety of buprenorphine transdermal patch (Norspan® patch 5 mg, 10 mg and 20mg) against oral tramadol (Tridol® SR (slow release) tablet 100mg) in patients with moderate to severe pain due to osteoarthritis.

DETAILED DESCRIPTION:
The primary objective of this non-inferiority study with active, parallel control group is to compare and assess efficacy and safety of buprenorphine transdermal patch (Norspan® Patch 5 mg, 10 mg and 20 mg) and tramadol (Tridol® SR (slow release) Tablet 100mg) in patients with moderate to severe pain due to osteoarthritis. During the period of treatment for 8weeks, titration and maintenance is kept up after 1:1 ratio randomization.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged more than 18 years.
* Clinical diagnosis of osteoarthritis (OA) of the hip and/or knee including fulfilling the American College of Rheumatology Criteria (ACR criteria L13) and documentation of osteoarthritis in the relevant joint.
* Patients with moderate to severe osteoarthritis pain in the relevant joint, confirmed by BS-11 (Box Scale-11) more than 4 for their pain on average during the last week, in their primary OA joint, at both the screening and base line visits despite treatment with non-opioid analgesics.

Exclusion Criteria:

* Patients being treated with high potency opioid analgesics (e.g., morphine, fentanyl, oxycodone, methadone, hydromorphone, ketobemidone, buprenorphine (including Norspan®)) for their osteoarthritis pain.
* Patients who have been taking any opioid analgesics within the last 4 weeks prior to the screening visit.
* Patients who have been using any (Non-steroidal Anti-Infammatory) NSAID transdermal preparation less than 2 weeks prior to the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Pain intensity - BS (box score)-11 pain scale | 8 weeks

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 8 weeks
Degree of sleep disturbance due to pain and improvement in quality of sleep | 8 weeks
Incidence of early discontinuation due to lack of efficacy | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Myun Chul Lee, Principal Investigator — Seoul National University Hospital
Locations (5):
- South Korea (5):
  - Asan Medical Center, Seoul
  - Hanyang University Medical Center, Seoul
  - National Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul